CLINICAL TRIAL: NCT02565342
Title: Interscalene Brachial Plexus Block to Treat Pain After Clavicular Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER 317/15
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Acute Pain
Keywords: Clavicle
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interscalene brachial plexus block (Experimental)
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block

SUMMARY:
The sensory innervation of the clavicle remains an area of debate. Regional nerve blocks aimed at relieving pre- and post-operative pain include the superficial cervical plexus blocks, interscalene blocks and a combined version of the above. In this case study, the investigators aim to describe the protocol used in a university hospital: general anaesthesia with interscalene brachial plexus block, followed by optional iv morphine administration in phase 1 recovery and oral oxycodone on the ward.

ELIGIBILITY:
Inclusion Criteria:

* clavicular fracture with internal reduction
* physical status I - III

Exclusion Criteria:

* contraindication to regional anaesthesia
* history of neck radiotherapy
* patient suffering from chronic pain
* severe respiratory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
IV Morphine consumption in phase 1 recovery (mg) | 0-2 hours after surgery
  morphine administered in postanaesthetic care unit by nursers if pains score > 3/10, per protocol

SECONDARY OUTCOMES:
Pain scores at rest and on movement (numeric rating scale, 0-10) | Postoperative day 0 and 1
Postoperative nausea and vomiting (yes/no) | Postoperative day 0 and 1
Itching (yes/no) | Postoperative day 0 and 1
Cumulative oxycodone consumption (mg) | up to postoperative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Olofsson M, Taffe P, Kirkham KR, Vauclair F, Morin B, Albrecht E. Interscalene brachial plexus block for surgical repair of clavicle fracture: a matched case-controlled study. BMC Anesthesiol. 2020 Apr 20;20(1):91. doi: 10.1186/s12871-020-01005-x. PMID 32312249